CLINICAL TRIAL: NCT05734261
Title: Interest of Forced Oscillations During a Methacholine Test in Children
Brief Title: Forced Oscillations Technique During a Metacholine Test in Children
Acronym: TPM AOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0504; 2022-A02437-36 (Other: ANSM); RECHMPL22_0504 (Other: CHU de Montpellier)
Record Dates: First submitted 2023-02-02; First posted 2023-02-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Asthma in Children
Keywords: Infant; Asthma; Diagnosis; Methacholin; Forced oscillation
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Intervention Model Description: Each subject is his or her own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other)
  Interventions: Procedure: Airway Oscillation System

INTERVENTIONS:
Procedure: Airway Oscillation System — After each methacholine dose administred, respiratory function will be measured by forced oscillation
  Other Names: Tremoflo

SUMMARY:
Asthma is the most common chronic lung disease in children. It affects more than 1 in 10 children in France. The methacholine bronchial challenge test (MBT) is indicated to assess the probability of asthma suggested by clinical symptoms by measuring the forced expiratory volume in one second (FEV1), after inhalation of a cumulative dose of methacholine. In children, the measurement of FEV1 requires a high level of cooperation from the child, which can be the source of false negatives or no result if this is not obtained. The objective of this study is to evaluate if the measurement of the respiratory function by the forced oscillations technique, allows to predict the variation of the FEV1 obtained

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 16 years
* FEV1 > 60%
* Child referred to the pulmonary function test laboratory for a non-specific bronchial hyperactivity test with methacholine
* Child under treatment with inhaled corticosteroids stopped for at least 3 weeks
* Oral consent from the child and at least one of the legal representatives
* Child affiliated or benefiting from a social security plan

Exclusion Criteria:

* Use of a short-acting beta-adrenergic bronchodilator within the last 6 hours or anticholinergic bronchodilator within the last 12 hours
* Use of a long-acting beta-adrenergic bronchodilator (licensed for use in children) in the past 36 hours
* Upper or lower respiratory tract infections within 3 weeks prior to inclusion
* Epilepsy under treatment
* Subject's participation in another interventional study that may alter respiratory function
* Patient unable to give consent, vulnerable

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in lung impedance measurement | During the procedure
  Percentage change in lung impedance measurement obtained by the forced oscillation technique in relation to the dose of methacholine required to obtain bronchial hyperresponsiveness

SECONDARY OUTCOMES:
Average number of trials required for measurement of FEV1 with the spirometry technique | During the procedure
  Average number of trials required for technically satisfactory iterative measurement of FEV1
Average number of trials required for impedance measurement by forced oscillation | During the procedure
  Average number of trials required for technically satisfactory iterative measurement of impedance

CONTACTS AND LOCATIONS:
Overall Officials: Stefan MATECKI, MD, Principal Investigator — Montpellier Univerty Hospital
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No